CLINICAL TRIAL: NCT04840485
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled, Phase II/III Adaptive Study of SHR-1314 to Assess Efficacy and Safety in Patients With Active Ankylosing Spondylitis
Brief Title: Efficacy and Safety of SHR-1314 in Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1314-302
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1314
- Treatment group B (Experimental)
  Interventions: Drug: SHR-1314
- Treatment group C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1314 — SHR-1314 high dose
  Arms: Treatment group A
Drug: SHR-1314 — SHR-1314 low-dose
  Arms: Treatment group B
Drug: Placebo — Placebo
  Arms: Treatment group C

SUMMARY:
The purpose of this study is to assess efficacy, safety, pharmacokinetics and immunogenicity of subcutaneous SHR-1314 in patients with active ankylosing spondylitis

ELIGIBILITY:
Inclusion Criteria:

- Active Ankylosing Spondylitis, prior radiographic evidence according to the Modified NY Criteria (1984), inadequate response, contraindications or intolerance to NSAIDs

Exclusion Criteria:

- pregnancy or lactation, serious infectious, malignancy, previous exposure to any biological agent excluding TNF antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Responded for Assessment of SpondyloArthritis international Society 20 Criteria (ASAS20) at 16 Weeks | 16 Weeks

SECONDARY OUTCOMES:
Percentage of Participants Responded for ASAS 20 Response at 32 Weeks | 32 Weeks
Percentage of Participants Responded for ASAS 40 Response at 16 and 32 Weeks | 16 and 32 Weeks
Percentage of Participants Responded for ASAS 5/6 Response at 16 and 32 Weeks | 16 and 32 Weeks
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at 16 and 32 Weeks | 16 and 32 Weeks
Change From Baseline in Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) at 16 and 32 Weeks | 16 and 32 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China